CLINICAL TRIAL: NCT03701061
Title: Human Immune Responses to an Adjuvanted H5 Vaccine: Durability and Impact of the Seasonal Influenza Vaccine on H5 Induced B Cell Response
Brief Title: Durability and Impact of the Seasonal Influenza Vaccine on H5 Induced B Cell Response
Acronym: HIPCVAX-010S
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Nadine Rouphael, Associate professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00100804; U19AI090023 (NIH)
Record Dates: First submitted 2018-10-06; First posted 2018-10-09 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Influenza A Subtype H5N1 Infection
Keywords: Immune response

STUDY DESIGN:
Intervention Model Description: Prospective, Exploratory study with up to 50 subjects total, who previously participated in the HIPCVAX-010 Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine with and without AS03 Adjuvant study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Participants that received AS03 Adjuvant (Experimental): Subjects that participated in HIPCVAX-010 Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine with AS03 Adjuvant study are included in the study. Subjects will receive a single dose of the FDA-approved 2018-2019 seasonal influenza vaccine (Fluarix Quadrivalent).
  Interventions: Biological: Seasonal Influenza Vaccine
- Participants that did not receive AS03 Adjuvant (Active Comparator): Subjects that participated in HIPCVAX-010 Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine without AS03 Adjuvant study are included in the study. Subjects will receive a single dose of the FDA-approved 2018-2019 seasonal influenza vaccine (Fluarix Quadrivalent).
  Interventions: Biological: Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Seasonal Influenza Vaccine — A single dose of the FDA-approved 2018-2019 seasonal influenza vaccine (Fluarix Quadrivalent) will be administered to the subjects participated in HIPCVAX-010 Study
  Other Names: Fluarix Quadrivalent
  Arms: Participants that received AS03 Adjuvant
Biological: Seasonal Influenza Vaccine — A single dose of the FDA-approved 2018-2019 seasonal influenza vaccine (Fluarix Quadrivalent) will be administered to the subjects participated in HIPCVAX-010 Study
  Other Names: Fluarix Quadrivalent
  Arms: Participants that did not receive AS03 Adjuvant

SUMMARY:
The study is a prospective single site exploratory study to examine the impact of Food and Drug Administration (FDA) approved seasonal flu vaccine on the immune responses of H5N1 vaccine previously received with or without the AS03 adjuvant.

DETAILED DESCRIPTION:
Influenza, caused by the influenza virus, is a contagious respiratory disease that can result in mild to severe illness. It is estimated that up to 80,000 deaths and approximately 200,000 Americans are hospitalized annually due to complications. Vaccination is the most effective way of controlling flu and preventing its illness and complications; however, antibody responses to seasonal influenza vaccines decrease over time and only target a small number of antibody binding sites In 2015, the Hope Clinic of the Emory Vaccine Center completed a study analyzing human immune responses to a pandemic H5N1, or "bird flu" vaccine, either alone or combined with the GlaxoSmithKline adjuvant system 03 (AS03).

Participants that took part in the 2013 HIPCVAX-010 Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine with and without AS03 Adjuvant study will be enrolled in this study to assess the effect of seasonal influenza vaccine in shaping the immune responses. The study aims to address important immunological mechanisms that can assist scientists in the creation of a universal influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Participated in HIPCVAX-010 Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine with and without AS03 Adjuvant study.
* Capable of informed consent and provision of written informed consent before any study procedures.
* Capable of attending all study visits according to the study schedule.
* Are in good health, as determined by medical history and targeted physical exam related to this history.
* Female subjects of childbearing age must have a negative urine pregnancy test before study vaccination, and must use at least one form of contraception to avoid pregnancy for 28 days before and 28 days after Fluarix Quadrivalent administration.

Exclusion Criteria:

* Have an acute illness, including any fever (> 100.4 F [> 38 degrees C], regardless of the route) within 72 hours before vaccination.
* Have any acute or chronic medical condition that, in the opinion of the principal investigator, would make vaccination unsafe or interfere with the evaluation of immune response to study vaccination.
* Alcohol or drug abuse and psychiatric conditions that, in the opinion of the investigator, would preclude compliance with the trial or interpretation of safety or endpoint data.
* Have a suppressed immune system as a result of illness, immunosuppressive medication, chemotherapy, or radiation therapy within 3 years prior to study vaccination.
* Are pregnant or breastfeeding or plan to within one month of vaccination.
* Have taken oral or parenteral corticosteroids of any dose within 28 days before study vaccination.
* Have a known history of autoimmune disease.
* Have a history of Guillain-Barre Syndrome.
* Have a history of bleeding disorders.
* Have known hypersensitivity or allergy to any component of the vaccine, including egg and latex allergies, or history of anaphylaxis with influenza vaccine or vaccine component.
* Have received blood or blood products 3 months prior to study entry or expected to receive through 6 months after study entry.
* Have received any live virus vaccines within 4 weeks prior to study entry or expected receipt within 4 weeks after study entry.
* Have received any inactivated vaccine within 2 weeks or expected receipt within 2 weeks after study entry.
* Have received any experimental agents within 6 weeks prior to study or plan to through study duration.
* Have received the 2018-2019 influenza seasonal vaccine.
* Documented influenza infection during the 2018-2019 influenza season.
* Social, occupational, or any other condition that in the opinion of the investigator might interfere with compliance with the study and vaccine evaluation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic of Emory University, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants That Received AS03 Adjuvant | Participants That Did Not Receive AS03 Adjuvant
Started | 9 | 3
Completed | 9 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants That Received AS03 Adjuvant: Subjects that participated in HIPCVAX-010 Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine with AS03 Adjuvant study (NCT01910519) are included in the study. Subjects will receive a single dose of the FDA-approved 2018-2019 seasonal influenza vaccine (Fluarix Quadrivalent).
  Seasonal Influenza Vaccine: A single dose of the FDA-approved 2018-2019 seasonal influenza vaccine (Fluarix Quadrivalent) will be administered to the subjects participated in HIPCVAX-010 Study
- Participants That Did Not Receive AS03 Adjuvant: Subjects that participated in HIPCVAX-010 Systems Biology of Influenza A (H5N1) Virus Monovalent Vaccine without AS03 Adjuvant study (NCT01910519) are included in the study. Subjects will receive a single dose of the FDA-approved 2018-2019 seasonal influenza vaccine (Fluarix Quadrivalent).
  Seasonal Influenza Vaccine: A single dose of the FDA-approved 2018-2019 seasonal influenza vaccine (Fluarix Quadrivalent) will be administered to the subjects participated in HIPCVAX-010 Study
- Total: Total of all reporting groups
Arm/Group | Participants That Received AS03 Adjuvant | Participants That Did Not Receive AS03 Adjuvant | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 3 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 2 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Four-fold Increase in Stem-specific Antibody Titers (H5, Hemagglutinin Antibody) Against H5N1 at Day 29 After Vaccination With the Seasonal Influenza Vaccine Among All the Participants in Both Arms
Description: Antibody Titers (hemagglutinin inhibition antibody titers) are measured through immunologic assays from blood draw at Baseline (Day1) before study vaccination and are repeated on Day 29. Participants with four fold increase in titer levels will be recorded.
Time Frame: Baseline (Day 1) before vaccination and Day 29 post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Participants That Received AS03 Adjuvant | Participants That Did Not Receive AS03 Adjuvant
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

2. Secondary Outcome: Number of Solicited (AE's) Grade 2 and Above at Day 8 After Vaccination With the Seasonal Influenza Vaccine Among the Participants in Both Arms
Description: To evaluate safety, grade 2 and above solicited AE's are recorded from Day 1 post vaccination to Day 8 post vaccination.Solicited adverse events include local (pain, erythema and induration) and systemic (chills, loss of appetite, headache, fatigue, myalgia, arthralgia, nausea, fever (body temperature ≥ 38°C (100.4°F)).
Time Frame: up to Day 8 post vaccination
Measure: Number; unit: number of events
Arm/Group | Participants That Received AS03 Adjuvant | Participants That Did Not Receive AS03 Adjuvant
Number analyzed (Participants) | 9 | 3
number of events | 1 | 0

3. Secondary Outcome: Number of Unsolicited Adverse Events (AE's) Grade 2 and Above at Day 29 After Vaccination With the Seasonal Influenza Vaccine Among the Participants in Both Arms
Description: To evaluate safety, grade 2 and above unsolicited AE's are recorded from Day 1 post vaccination to Day 29 post vaccination. Unsolicited AE information is volunteered or noted in an unsolicited manner and not as a required data element through a case report form.
Time Frame: Up to Day 29 post vaccination
Measure: Number; unit: number of events
Arm/Group | Participants That Received AS03 Adjuvant | Participants That Did Not Receive AS03 Adjuvant
Number analyzed (Participants) | 9 | 3
number of events | 0 | 0

4. Secondary Outcome: Number of Serious Adverse Events at Day 365 Among the Participants in Both Arms
Description: Serious adverse events are recorded from Day 1 post vaccination to Day 365 post vaccination. A serious adverse event is any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, or is considered an "other important medical event" based on medical judgement.
Time Frame: Up to 365 days post vaccination
Measure: Number; unit: number of events
Arm/Group | Participants That Received AS03 Adjuvant | Participants That Did Not Receive AS03 Adjuvant
Number analyzed (Participants) | 9 | 3
number of events | 0 | 0

ADVERSE EVENTS:
Time Frame: from Day 1 post vaccination to Day 365 post vaccination
Arm/Group | Participants That Received AS03 Adjuvant | Participants That Did Not Receive AS03 Adjuvant
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 1/9 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants That Received AS03 Adjuvant (N=9) | Participants That Did Not Receive AS03 Adjuvant (N=3)
Headache (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT03701061/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03701061/Prot_SAP_001.pdf